CLINICAL TRIAL: NCT05374720
Title: Analysis of the Molecular Composition of Tubal Cilia in Patients With or Without Ectopic Pregnancy
Acronym: CILTUBE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CILTUBE
Record Dates: First submitted 2022-03-07; First posted 2022-05-16 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Salpingectomy; Hysterectomy; Primary Ciliary Dyskinesia; Ectopic Pregnancy
Keywords: miscarriage; tubal cilia
MeSH Terms: conditions — Ciliary Motility Disorders; Pregnancy, Ectopic; Abortion, Spontaneous | interventions — Salpingectomy; Hysterectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salpingectomy for Extra-Uterine Pregnancy (Experimental): patients with salpingectomy for Ectopic Pregnancy
  Interventions: Procedure: salpingectomy
- hysterectomies (Sham Comparator): patients with hysterectomy for prolapsus, adenomyosis or myomectomy
  Interventions: Procedure: hysterectomy

INTERVENTIONS:
Procedure: salpingectomy — Removal of one of the fallopian tubes.
  Arms: Salpingectomy for Extra-Uterine Pregnancy
Procedure: hysterectomy — remove the uterus, whole or only part. It may also involve the removal of the cervix, ovaries, fallopian tubes and other surrounding structures.
  Arms: hysterectomies

SUMMARY:
Primary Ciliary Dyskinesia associated with abnormalities of lateralization of organs (with existence of a situs inversus in 50% of cases) and secondary fertility disorders related in humans to abnormalities of mobility of sperm but very little data on the structure and function of tubal cilia in women

DETAILED DESCRIPTION:
Primary Ciliary Dyskinesia (DCP) is a rare genetic disease (1 in 15,000 individuals at birth), which manifests itself in chronic respiratory infections (bronchopneumopathies and rhinosinusitis type) associated with abnormalities of lateralization of organs (with existence of a situs inversus in 50% of cases) and secondary fertility disorders related in humans to abnormalities of sperm mobility. However, there is very little data in the literature on the structure and function of tubal cilia in women with DCP.

Before considering a study of tubal cilia in patients with DCP, it seems necessary to specify in DCP patients or not DCP, the molecular and morphological composition of tubal cilia and to look for ciliary abnormalities in case of GEU

ELIGIBILITY:
Inclusion Criteria:

* Patients with scheduled salpingectomy (Ectopic pregnancy, hysterectomy for prolapsus, adenomyosis or myomectomy)
* Major patients ( >18 years)

Exclusion Criteria:

* Patient not willing to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
morphological of tubal cilia | through study completion, an average of 6 week after surgery
  Molecular compositor of tubal ciliar by immunofluorescence study of 14 proteins in vivo and in vitro (tissue cells from patient fallopian tubes)
Molecular difference in tubal cilia between patients with or without GEU salpingectomy | through study completion, an average of 6 week after surgery
  compares molecular compositor of tubal ciliar by immunofluorecence study of 14 proteins in vivo and in vitro between patients with or without GEU salpingectomy
molecular tubal cilia | through study completion, an average of 6 week after surgery
  Ultrastructure morphology of tubal cell cilia by electron microscopy
functional composition of tubal cell by video microscopy | through study completion, an average of 6 week after surgery
  amplitude of moment by video microscopy
functional composition of tubal cell by video microscopy | through study completion, an average of 6 week after surgery
  frequency of moment by video microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Rana i MITRI-FRANGIEH, Principal Investigator — Centre Hospitalier Intercommunal Créteil
Locations (1):
- Centre Hospitalier Intercommunal Créteil, Créteil, Val-deMarne, France